CLINICAL TRIAL: NCT06132178
Title: Assessing the Safety, Tolerability, and Efficacy of Psilocybin Therapy Followed by Accelerated Intermittent Theta Burst (aiTBS) Repetitive Transcranial Magnetic Stimulation (rTMS) for Treatment-Resistant Major Depressive Disorder
Brief Title: Psilocybin rTMS for Treatment Resistant Depression
Acronym: PSILOBSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Greg Fonzo, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004537
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Treatment Resistant Depression; MDD; Major Depressive Disorder; Recurrent Depression; Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depression | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This will be a phase II 2x2 design (device and dose) clinical trial. 100 participants, ages 22-76, with treatment-resistant MDD will be randomized to treatment with either: a) 25mg of COMP360 (N=50); or b) 1mg of COMP360 (low-dose comparator; N=50) with appropriate psychological preparation, support, and integration sessions with trained therapists. This will then be directly followed by one of two subsequent treatment conditions: i) the active accelerated intermittent theta burst (aiTBS) rTMS treatment known as Stanford Neuromodulation Therapy (SNT) and/or Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) targeted to a functional magnetic resonance imaging (fMRI) functional connectivity-guided personalized left dorsolateral prefrontal cortex target using neuronavigation and delivered over 10 sessions daily for 5 consecutive days at 90% of coil-to-target depth-corrected resting motor threshold50,51; or ii) sham iTBS delivered in the same fashion.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Full dose COMP360 with active aiTBS rTMS (Experimental): 25mg of COMP360 with the active accelerated intermittent theta burst (aiTBS) rTMS treatment known as Stanford Neuromodulation Therapy (SNT) and/or Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) delivered over 10 sessions daily for 5 consecutive days.
  Interventions: Drug: Psilocybin; Device: Accelerated intermittent theta burst (aiTBS) rTMS treatment
- Full dose COMP360 with sham aiTBS rTMS (Active Comparator): 25mg of COMP360 with sham iTBS delivered over 10 sessions daily for 5 consecutive days.
  Interventions: Drug: Psilocybin; Device: Sham Accelerated intermittent theta burst (aiTBS) rTMS treatment
- Low dose comparator with active aiTBS rTMS (Active Comparator): 1mg of COMP360 with the active accelerated intermittent theta burst (aiTBS) rTMS treatment known as Stanford Neuromodulation Therapy (SNT) and/or Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) delivered over 10 sessions daily for 5 consecutive days.
  Interventions: Device: Accelerated intermittent theta burst (aiTBS) rTMS treatment; Drug: Low-dose psilocybin
- Low dose comparator with sham aiTBS rTMS (Sham Comparator): 1mg of COMP360 with with sham iTBS delivered over 10 sessions daily for 5 consecutive days.
  Interventions: Drug: Low-dose psilocybin; Device: Sham Accelerated intermittent theta burst (aiTBS) rTMS treatment

INTERVENTIONS:
Drug: Psilocybin — A psychedelic drug found in certain mushrooms. It will be in a capsule of 25mg psilocybin (COMP360).
  Other Names: COMP360
  Arms: Full dose COMP360 with active aiTBS rTMS; Full dose COMP360 with sham aiTBS rTMS
Device: Accelerated intermittent theta burst (aiTBS) rTMS treatment — A form of non-invasive brain stimulation that delivers a series of quick magnetic pulses to the scalp and a portion of the brain. It will be targeted to a functional magnetic resonance imaging (fMRI) functional connectivity-guided personalized left dorsolateral prefrontal cortex target using neuronavigation and delivered over 10 sessions daily for 5 consecutive days at 90% of coil-to-target depth-corrected resting motor threshold.
  Other Names: Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT); Stanford Neuromodulation Therapy (SNT)
  Arms: Full dose COMP360 with active aiTBS rTMS; Low dose comparator with active aiTBS rTMS
Drug: Low-dose psilocybin — A psychedelic drug found in certain mushrooms. It will be in a low-dose form of the experimental dose as a 1mg capsule of psilocybin (COMP360).
  Other Names: low-dose COMP360
  Arms: Low dose comparator with active aiTBS rTMS; Low dose comparator with sham aiTBS rTMS
Device: Sham Accelerated intermittent theta burst (aiTBS) rTMS treatment — The sham version is meant to look and feel like the active SAINT rTMS, but the main difference is that the brain is not being stimulated like the active condition.
  Other Names: Sham Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT); Sham Stanford Neuromodulation Therapy (SNT)
  Arms: Full dose COMP360 with sham aiTBS rTMS; Low dose comparator with sham aiTBS rTMS

SUMMARY:
The purpose of this study is to determine the safety and feasibility of sequencing psilocybin therapy with a short-duration, aiTBS protocol (Stanford Accelerated Intelligent Neuromodulation Therapy, or SAINT) in individuals with treatment-resistant major depressive disorder.

DETAILED DESCRIPTION:
This will be a phase II 2x2 design (device and dose) clinical trial. 100 participants, ages 22-76, with treatment-resistant MDD will be randomized to treatment with either: a) 25mg of COMP360 (N=50); or b) 1mg of COMP360 (low-dose comparator; N=50) with appropriate psychological preparation, support, and integration sessions with trained therapists. This will then be directly followed by one of two subsequent treatment conditions: i) the active accelerated intermittent theta burst (aiTBS) rTMS treatment known as Stanford Neuromodulation Therapy (SNT) and/or Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT) targeted to a functional magnetic resonance imaging (fMRI) functional connectivity-guided personalized left dorsolateral prefrontal cortex target using neuronavigation and delivered over 10 sessions daily for 5 consecutive days at 90% of coil-to-target depth-corrected resting motor threshold50,51; or ii) sham iTBS delivered in the same fashion. Individuals will undergo screening, a baseline clinical assessment and neurobiological assessment of functional magnetic resonance imaging (fMRI) and electroencephalographic (EEG) recordings. Individuals will then return on a subsequent day to begin the course of psilocybin therapy. Preparation sessions will occur on the first two out of five days (~1.5-2 hrs each day), psilocybin dosing will occur on the third day (~6-8 hours), integration session (~1 hour) and post-dosing assessments will occur on the fourth day, and a final integration session (~1 hour) and post-psilocybin clinical and neurobiological assessments will occur on the last of the five days. The following week, the individual will return to the lab to begin the course of active or sham SNT, for 10 hrs. a day (10 min once per 60 min, 50-minute inter-session interval, repeated 10 times daily) for 5 days. This is the protocol now FDA-cleared for treatment of treatment-resistant MDD, known as Stanford Neuromodulation Therapy and commercialized by Magnus Medical (see support letter from Magus Medical). In the third week, the individual will return to complete post-SNT clinical assessments and to complete a post-SNT neurobiological (fMRI and EEG) assessment. Individuals will complete long-term follow-up clinical assessments at 1 month, 2 months, 3 months, 4 months, 6 months, 9 months, and 12 months post-initiation of first treatment (psilocybin administration) to assess durability of clinical response and identify potential points of depression relapse over a sustained period of time.

Aims:

To determine the safety and feasibility of sequencing psilocybin therapy with a short-duration, aiTBS protocol (Stanford Accelerated Intelligent Neuromodulation Therapy, or SAINT) in individuals with treatment-resistant major depressive disorder.

To determine if the combination of psilocybin therapy followed by SAINT demonstrates superior efficacy relative to either treatment alone acutely (primary acute endpoint will be ~14 days after the initiation of the treatment sequence) and over time (additional endpoints at 2 weeks, 4 weeks, 2 months, 3 months, 4 months, 5 months, 6 months, 9 months, and 12 months following cessation of the treatment protocol).

To determine the neurobiological changes following the combination treatment (assessment points at baseline, 2 days post-psilocybin, and ~14 days post-psilocybin/2-4 days post cessation of accelerated theta burst), and if the magnitude or nature of such changes are different from those demonstrated in either treatment alone.

Investigate how psychedelic treatment may impact blood biomarkers of inflammation (e.g., inflammatory cytokines) and how select functional genetic polymorphisms may moderate the effect of the psychedelic treatment on subsequent functional brain changes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, ages 22-65.
2. English language comprehension suitable to understand experimenter instructions and to communicate to study personnel/staff reasonably easily.
3. Current major depressive episode (without psychotic features), either as part of recurrent major depressive disorder (MDD) or single episode MDD with current episode present for at least the past 3 months (as determined by the Structured Clinical Interview for DSM-5; SCID-5).
4. Montgomery Asberg Depression Rating Scale (MADRS) score of 20 or greater at baseline assessment (at least moderate severity).
5. 1. Treatment-resistant MDD, defined as either: a) failure to respond to an adequate dose and duration of two or more pharmacological treatments, with at least one failed medication trial occurring in the current major depressive episode; or b) failure to respond to an adequate dose and duration of 2 or more pharmacological treatments of different pharmacological classes in one or more past major depressive episodes. Adequate treatment dose and duration will be determined through the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ). Augmentation, where an add-on medication is used, will be counted as a second treatment, provided it is approved as an adjunctive treatment of MDD in the country where prescribed.
6. Willingness and ability to attend daily, full-day visits to the research site for a period of ~2 weeks and to participate in all study procedures (clinical assessments, treatments, and neurobiological assessments).
7. If currently taking an antidepressant medication (an SSRI, SNRI, or atypical antidepressant), antipsychotic, and/or other augmenting medication (e.g., lithium), willingness to discontinue medication(s) over a 2-8 week period with the assistance of study staff and maintain at least a 2-5 week period (5-week period for fluoxetine) off of medications prior to the baseline visit AND willingness to remain off medications for a period of 1 month following the end of the treatment course (approximately 6-8 weeks after the baseline visit).

Exclusion Criteria:

1. Prior history or current diagnosis of a psychotic disorder (including MDD with psychotic features), bipolar disorder, or personality disorder (based on medical history, clinician judgement, SCID-5 and/or SCID for Personality Disorders).
2. Current diagnosis of posttraumatic stress disorder, acute stress disorder, obsessive-compulsive disorder, anorexia nervosa, bulimia nervosa, or alcohol or substance-use disorder.
3. Having met criteria for an alcohol or substance-use disorder within the past year.
4. Use of electroconvulsive therapy, deep brain stimulation, or vagus nerve stimulation during the current major depressive episode.
5. Any prior rTMS treatment (10Hz, 5Hz, 1Hz, or conventional intermittent theta burst).
6. Current participation in an evidence-based psychotherapy for major depression (e.g., cognitive behavioral therapy, behavioral activation). Ongoing supportive psychotherapy is allowable if maintained at the same frequency throughout the duration of the short-term follow-up clinical endpoint (1 month after treatment cessation) of the study and if no recent change in therapy type or frequency for 1 month prior to enrollment.
7. Exhibiting significant suicide risk within the past 12 months, at screening, or at baseline, as evidenced by: a) suicidal ideation with some intent to act but no specific plan (item #4 from the Columbia Suicide Severity Rating Scale57; C-SSRS); b) suicidal ideation with intent to act and a specific plan (item #5 from the C-SSRS); c) suicide attempt or non-suicidal self-injury requiring medical attention in the past 12 months; or d) self-report of significant suicidal ideation with intent or significant non-suicidal self-injury during screening or baseline clinical interview.
8. Major depressive episode that is secondary to a medication or a general medical condition, as judged by investigators.
9. Any other factors, such as major medical conditions, unstable housing or threatening life circumstances, erratic behavior, etc. that are judged by the investigators to be a significant barrier to participation in the study protocol and/or to establishing therapeutic rapport necessary for safe administration of psilocybin.
10. Prior past-year ingestion of a serotonergic psychedelic, e.g., psilocybin, LSD, mescaline, dimethyltryptamine, etc. or more than 5 lifetime ingestions of a serotonergic psychedelic on separate occasions.
11. Participant unwillingness to not ingest or use additional serotonergic psychedelics outside the context of study procedures for the duration of the study follow-up period (12 months).
12. Ferrous metal, metallic implants, or implanted medical devices that would preclude administration of rTMS and/or participation in MRI procedures, including but not limited to: cochlear implants, implanted brain stimulators, aneurysm clips.
13. Past history of seizures or epilepsy (rTMS risk).
14. Neurological disorder, including epilepsy, stroke, or history of brain surgery.
15. Past penetrating brain injury or any head injury resulting in a loss of consciousness for 30 minutes or more or post-concussive symptoms for more than seven days following a head injury.
16. Head injury in the past two months, regardless of severity.
17. Currently pregnant and/or nursing or about to become pregnant. A positive urine pregnancy test at screening and/or baseline will lead to participant exclusion from the study.
18. Engagement in sexual intercourse which could result in pregnancy without use of a highly effective contraceptive method throughout participation in the study and for at least three months after COMP360 (psilocybin) administration.
19. Severe claustrophobia (prohibiting MRI acquisition).
20. Uncontrolled hypertension (resting blood pressure > 140/90 mm hg).
21. Uncontrolled thyroid disease as indicated by unstable thyroid hormone dosage < 3 months prior to screening, or abnormal and clinically significant thyroxine (FT4) levels (a free FT4 measurement will be conducted for all participants with an out-of-range thyroid-stimulating hormone [TSH] value irrespective of thyroid history).
22. Lifetime history of cardiomyopathy, stroke, heart disease, heart attack, tachycardia, elongated QT-interval corrected by Friderichia (> 450ms for men and > 470ms for women); clinically significant cardiac arrhythmia within 1 year of study entry; and/or abnormal electrocardiogram on study entry.
23. Type I diabetes mellitus or uncontrolled Type II diabetes mellitus (defined by hemoglobin A1c > 8% at screening) or a history of diabetic ketoacidosis, hyperglycemic coma, or severe hypoglycemia with loss of consciousness (< 3 months prior to signing of consent form).
24. Positive urine drug screening for drugs of abuse at screening and/or baseline will trigger a review with participant and assessment for eligibility based on pattern of use and willingness to abstain in conjunction with medical monitor and investigative team.
25. Clinically-significant results from physical examination, blood test, urine test, vital signs, or ECG at screening and/or baseline.
26. Current enrollment in another interventional study or participation within such a study within 6 months of screening.
27. Self-reported hypersensitivity to psilocybin or another serotonergic psychedelic.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 12 months
  A ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Scoring ranging from 0 to 60, with higher scores indicating greater depressive symptomology.
fMRI task-evoked brain activation | At both 1 week and 2 weeks
  A method used in functional magnetic resonance imaging (fMRI) to observe different areas of the brain or other organs, which are found to be active at any given time.
fMRI resting state | At both 1 week and 2 weeks
  A method aimed at examining intrinsic networks in the brain while no task is performed (rest) in order to estimate correlations between brain regions.
EEG functional connectivity change | At both 1 week and 2 weeks
  A method aimed at examining intrinsic networks in the brain to estimate correlations between brain regions.

SECONDARY OUTCOMES:
Snaith Hamilton Pleasure Scale (SHAPS) | 12 months
  A self-report measure of anhedonia. Scoring range from 0 to 14, with lower scores indicating less anhedonia.
Quick Inventory of Depressive Symptom Self-Report (QIDS-SR) | 12 months
  A self report measure of depressive symptoms. Scores range from 0 to 48, with lower scores indicating less symptoms of depression.
World Health Organization Quality of Life Inventory-Brief subscale (WHO-QL-Brief) | 12 months
  A self-report measure of quality of life with four subscales: Physical Health, Psychological Health, Social Relationships, and Environment. Scores for each range from 4-20, with higher scores indicating better quality of life.
Beck Depression Inventory II (BDI II) | 12 months
  A self-report measure of positive and negative affect. There are scores for Positive Affect and Negative Affect, each of which is scored from 10-50. Higher scores indicate more of that particular type of affect.
Anxiety Sensitivity Index 3 (ASI-3) | 12 months
  A self-report measure of anxiety sensitivity. Scores range from 0 to 72, with lower scores indicating less anxiety sensitivity.
Beck Anxiety Inventory (BAI) | 12 months
  A self report measure of anxiety symptoms. Scores range from 0 to 63, with lower scores indicating less anxiety.
Mood and Anxiety Symptom Questionnaire 30 item Anhedonic Depression subscale (MASQ-30) | 12 months
  A subscale measure of anhedonic depressive symptoms. Scores range from 10-50, with lower scores indicating less anhedonic depression.
Mood and Anxiety Symptom Questionnaire 30 item Anxious Arousal subscale (MASQ-30) | 12 months
  A subscale measure of anxious arousal symptoms. Scores range from 10-50, with lower scores indicating less anxious arousal.
Physicians Health Questionnaire 9 (PHQ-9) | 12 months
  A self-report screener of major depression. Scores range from 0 to 27, with lower scores indicating fewer symptoms of depression.
Generalized Anxiety Disorder 7 (GAD-7) | 12 months
  A self-report screener of generalized anxiety disorder. Scores range from 0 to 21, with lower scores indicating less symptoms of generalized anxiety.
Columbia-Suicide Severity Rating Scale (C-SSRS) | 12 months
  Clinician-administered measure of suicidal ideation. Scores range from 0 to 25, with higher scores indicating more severe suicidal ideation.
Anger Attacks Questionnaire (AAQ) | 12 months
  Self-report measure of anger outbursts. Scores range from 5-25, with higher scores indicating more severe expressions of anger.
Brief Psychiatric Rating Scale (BPRS) | 2 weeks
  A tool clinicians or researchers use to measure psychiatric symptoms such as anxiety, depression, and psychoses. Scores range from 18 to 126, with lower scores indicating less severe psychiatric symptoms a score of 18 meaning no symptoms present.
Sheehan Disability Scale (SDS) | 12 months
  Self-report screener that measures impairment in functioning and generates 4 scores: a work disability score, a social life disability score, a family life disability score and a total score. To get a total score add up the 3 individual scores (work: social life: family life). The maximum possible score is 30, meaning more severe impairment from experienced disability.
Positive and Negative Affect Scale Short Form (PANAS-SF) | 12 months
  Self-Report scale that consists of different words that describe feelings and emotions to measure positive and negative affect. Scores are divided into two categories: 1) can range from 10-50 with higher scores representing higher levels of positive affect and 2) can range from 10-50 with lower scores representing lower levels of negative affect.
Acceptance and Action Questionnaire II (AAQ II) | 12 months
  Self-report measure that tracks how individuals are applying flexibility skills to their daily lives. 7 item scale with scores ranging from 7-49,with higher scores indicating higher psychological inflexibility, experiential avoidance, and more potential for psychological stress.
NEO Five Factor Inventory (NEO-FFI) | 12 months
  Self-report measure that assesses subjects for five domains of normal personality: neuroticism, extraversion, conscientiousness, agreeableness, and openness. Each domain is a 12-item scale with scores ranging from 12-60 where the combined scores create a personality profile.
Emotion Regulation Questionnaire (ERQ) | 12 months
  A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Assesses cognitive reappraisal (6 items) and expressive suppression (4 items) on a 7-point Likert-type response scale, with higher scores on each scale indicate greater use of the corresponding emotional regulation strategy. Min 10 - max 70.
UCLA Loneliness Scale 3 (UCLA-LS-3) | 12 months
  Clinician administered scale that comprises 3 questions that measure three dimensions of loneliness: relational connectedness, social connectedness, and self-perceived isolation. Each item is rated on a 3-point scale for a range of 3-9, with higher scores meaning more intense feelings of the 3 dimensions of loneliness.
Freiberg Mindfulness Inventory (FMI) | 12 months
  Self-report questionnaire for measuring mindfulness. A 14-item scale with scores 14-56 with higher scores meaning a higher degree of mindfulness.
Discontinuation Emergent Signs and Symptoms Scale | 1 week
  Self-report measure of 43-items that assess changes in symptomology when starting a new treatment. This measures does not correlate scores to an outcome but is used to assess the development of a new symptom or the worsening of an already existing one.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Fonzo, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- Health Discovery Building (HDB), 1601 Trinity St., Bldg B., Z0600, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
If participants chose to, they can be included in the Department of Psychiatry's Registry (Protocol 2020-04-0046). Participants may elect to be part of this registry, but this is not required as part of the participation in the current study. No other plans for sharing data outside of a research related inquiry for research purposes is expected. The registry informed consent will be provided to the participant if interested and consent will be obtained per procedures outlined in the registry protocol. De-identified data may be shared with future researchers for scientific purposes. If our lab shares biospecimens with future researchers, it will only be de-identified data. In this case, it will be shared in the form of an aggregated database with no PHI or PII included.